CLINICAL TRIAL: NCT06439667
Title: Virtually Supervised Tele-Exercise Platform for Accelerating Plantar Wound Healing
Brief Title: Tele-Exercise Platform for Plantar Wound Healing
Acronym: Tele-FootX
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: BioSensics (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor of Surgery, University of California, Los Angeles
Other Study IDs: IRB-24-6284; 1R43AG082614-01 (NIH)
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Ulcer; Wound Healing; Wound Care
Keywords: Diabetic Foot Ulcer; Ambulatory in the home without the aid of another person; Able to provide written informed consent
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is design and use a telemedicine platform which integrates video-chat, pre-programmed interactive game-based foot, and ankle exercise modules, and real-time quantitative performance metrics displayed to the clinician to improve patient's perfusion to the lower extremity, improve diabetic wound healing and prevent muscle loss in the lower extremity.This is a cross sectional and comparative feasibility study. It is designed to explore acceptability, feasibility and proof of concept/ .

DETAILED DESCRIPTION:
Foot ulceration is the most common and costly late complication of diabetes, with morbidity and mortality being worse than many cancers. It is estimated that up to one-third of people with diabetes will develop a diabetic foot ulcer (DFU) in their lifetime. Non-healing DFUs are a leading cause of hospitalization, amputation, disability, and death among people with diabetes. In the United States, one-third of all diabetes-related costs are spent on diabetic foot care, with two-thirds of the costs incurred in inpatient settings, constituting a substantial economic burden to society. Therefore, every means possible should be used to try to heal DFU and prevent amputation. In this regard, there is a significant body of evidence related to the clinical benefits of exercise for people with DFU, including improving blood flow and oxygen supply, muscle loss prevention, and joint mobility. Despite this evidence, exercise is not part of the standard care for wound healing, mainly because there is no solution for promoting and managing home-based exercise programs for people with DFU.

To address the gaps described above, the investigators propose an interactive foot and ankle tele-exercise platform called "Tele-FootX". This platform allows clinicians to remotely and virtually supervise exercise tasks and coach patients to perform evidence-based foot and ankle exercises inspired by the validated Buerger-Allen (BA), while also educating and monitoring the patients adherence to the exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults (age 18 years and older)
* Having Diabetic foot ulcer
* Ambulatory (in the home without the aid of another person)
* Willing and able to provide informed consent

Exclusion Criteria:

* Foot wound present for more than a year
* HbA1c > 12%
* ABI index limb is <0.60 and/or they are being considered for revascularization within the course of the study
* Ulcer involving bone or tendon
* Ulcer not caused by diabetes
* Fully confined to a wheelchair
* Any condition limiting the ability to engage in Tele-FootX exercise routine such as major cognitive decline, and major visual or hearing problem
* Unable or unwilling to attend prescribed clinic visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Convenient and selected based on available resources to demonstrate feasibility and the proof of concept effectiveness.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Tissue Oxygen Saturation (SatO2) | baseline, 15 minutes
  For measuring tissue oxygen saturation (SatO₂), we will use a validated, non-invasive near-infrared (NIR) imaging device (Snapshot NIR, KENT Imaging Inc., Calgary, AB, Canada). The device estimates SatO₂ levels in superficial tissue by tracing the wound perimeter in real-time. To minimize bias related to wound size and SatO₂ measurement, all wounds will be traced along their internal borders-excluding surrounding skin-using a standardized technique across all participants. Measurements will be conducted at baseline and at the end of the Tele-FootX session, which is expected to last approximately 15 minutes.

SECONDARY OUTCOMES:
Muscle Activation | 15 minutes
  To assess muscle activation and fatigue in response to each exercise program, surface electromyography (sEMG) sensors will be placed on the tibialis anterior and gastrocnemius muscles. Muscle fatigue will be evaluated by analyzing the power spectrum of sEMG signals using the Welch Periodogram. Measurements will be taken during the first and last minutes of the continuous, interactive Tele-FootX session. Mean frequencies and amplitudes will be compared between these intervals to assess fatigue. We anticipate no significant change in amplitude or frequency, indicating minimal to no muscle fatigue.
Percentage of successfully completed leg exercise tasks within a 10-Minute session | 10 minutes
  Feasibility will be assessed by evaluating participants' ability to complete all prescribed exercise tasks as guided by the Tele-FootX and Buerger-Allen exercise programs, each designed to be completed within a 10-minute session. Feasibility will be quantified as the percentage of successfully completed tasks, defined as exercises performed with sufficient angular velocity or range of motion, based on predefined thresholds. This percentage is calculated by dividing the number of successfully completed tasks by the total number of prescribed tasks within the session.

CONTACTS AND LOCATIONS:
Locations (1):
- University California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is an NIH SBIR study with a subaward from BioSensics. According to the contract agreement, any sharing of individual-level data may require prior approval from BioSensics, particularly if the data is intended for commercial or for-profit use.

REFERENCES:
- [Background] Finco MG, Najafi B, Zhou H, Hamad A, Ibrahim R, Al-Ali F. Game-based intradialytic non-weight-bearing exercise training on gait speed and balance in older adults with diabetes: a single-blind randomized controlled trial. Sci Rep. 2023 Aug 30;13(1):14225. doi: 10.1038/s41598-023-41290-3. PMID 37648695
- [Background] Lee M, Hamad A, Azarian M, Beom J, Ouattas A, Dehghan Rouzi M, Rodriguez N, Quach N, Ibrahim R, Mathew M, Talal T, Al-Ali F, Najafi B. Efficacy and Feasibility of Intradialytic Plantar Electrical Stimulation in Patients With Diabetes: A Randomized Double-Blind Controlled Trial. Diabetes Care. 2024 Dec 1;47(12):2205-2213. doi: 10.2337/dc24-0928. PMID 39316389